CLINICAL TRIAL: NCT03611166
Title: iTRAQ-Based Proteomics Reveals Potential Biomarkers for Chronic Disorder of Consciousness
Brief Title: Proteomics for Chronic Disorder of Consciousness
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: proteomics
Record Dates: First submitted 2018-03-18; First posted 2018-08-02 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2017-12

CONDITIONS: Disorder of Consciousness
Keywords: proteomics; plasma; chronic disorder of consciousness
MeSH Terms: conditions — Consciousness Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood (5 mL) was collected in a Vacutainer® tube, containing anticoagulant, using standardized phlebotomy procedures. Plasma was prepared by centrifugation (2,000 g, 5 min, 4°C) and stored at -80°C until further analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Following severe traumatic brain injury, patients may remain unconscious for many years. It is the first proteomic analysis comparing differentially expressed proteins between patients with chronic disorder of consciousness and controls so far. The investigators generated accurate lists of proteomes and identified differences at different disease time courses. The obtained results provide new insight into understanding the molecular mechanisms underlying the chronic disorder of consciousness.

DETAILED DESCRIPTION:
Background: Patients who awake from severely traumatic brain injury (sTBI) may remain unconscious for many years. Although behavioral assessment and functional imaging are currently used as diagnostic tools, the molecular basis underlying chronic condition has yet to be explored.

Objective:To explore the molecular basis and identify novel biomarkers for the diagnosis and prognosis of patients with chronic disorder of consciousness.

Method: Plasma samples were obtained from patients with chronic disorder of consciousness, and healthy volunteers. A coupled isobaric tag for relative and absolute quantitation (iTRAQ)-based proteomics approach was used to screen differentially expressed proteins (DEPs) between patients and controls. Potential molecular mechanisms were further discussed through bioinformatics analyses. Candidate proteins were validated by enzyme-linked immunosorbent assay (ELISA).

ELIGIBILITY:
Inclusion Criteria:

1. Patients ages 14 to 65 years old;
2. Patients had a history of sTBI;
3. Patients had awakened from a coma (indicating preserved sleep-wake cycles), including vegetative state and minimally consciousness state;
4. Patients stay unconscious for more than 1 month.

Exclusion Criteria:

1. Patients with acute infectious diseases or liver dysfunction;
2. Patients with serious diseases such as cardiac or pulmonary problems.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with chronic disorder of consciousness were recruited at the rehabilitation units of Hangzhou Wujing Hospital (Hangzhou, Zhejiang, China).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-11-01 (Actual); Primary Completion 2019-06-15 (Estimated); Study Completion 2020-01-15 (Estimated)

PRIMARY OUTCOMES:
Protein profiling | Three months
  A coupled isobaric tag for relative and absolute quantitation (iTRAQ)-based proteomics approach was used to screen differentially expressed proteins (DEPs) between patients and controls.

SECONDARY OUTCOMES:
Glasgow Outcome Scale (GOS) | In one year
  A GOS value of <3 was considered as a bad recovery, while a GOS value of ≥3 was considered as a good recovery.
Coma Recovery Scale-Revised(CRS-R) | 30 minutes before blood collection
  Coma Recovery Scale-Revised (CRS-R) score was used to quantify the severity, which consists of 23 hierarchically arranged items that comprise six subscales addressing auditory, visual, motor, oromotor/verbal, communication, and arousal processes. The lowest item on each subscale represents reflexive activity, whereas the highest items represent cognitively mediated behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Benyan Luo, PHD, Principal Investigator — Department of Neurology and Brain Medical Centre The First Affiliated Hospital, School of Medicine, Zhejiang University 79 Qingchun Road, Hangzhou; Jian Gao, Principal Investigator — Hangzhou Hospital of Zhejiang CAPR,Hangzhou, Zhejiang, China; Hai Zou, Principal Investigator — Department of Cardiology, Zhejiang Provincial People's Hospital, Hangzhou, PR China
Locations (1):
- Hangzhou Hospital of Zhejiang CAPR, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No